CLINICAL TRIAL: NCT07108348
Title: The Effect of ADAR1 Expression Level on Total Neoadjuvant Treatment Response in Locally Advanced Rectal Cancer
Brief Title: ADAR1 Expression Level in Rectal Cancer
Acronym: ADAR1TNT
Status: Recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Turkish Society of Medical Oncology (Unknown)
Responsible Party: Principal Investigator, Mehmet Artac, MD, Necmettin Erbakan University
Other Study IDs: 24948/2025/5785; Turkish Society of Med. Onc. (Other: Turkish Society of Medical Oncology)
Record Dates: First submitted 2025-07-01; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Rectum Cancer, Adenocarcinoma
Keywords: ADAR1; rectum cancer; TNT
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Total RNA will be isolated from tissue samples stored at -80°C. In this process, 5-30 mg of tissue will be homogenized in a 1.5 mL homogenization tube, and then the extraction process will be performed according to the kit manufacturer's instructions, resulting in 30-50 μl of Total RNA. cDNA will be obtained from the RNA samples whose quantities have been calculated. In the PCR protocol, primer binding will be performed at 25°C for 10 minutes, reverse transcription will be performed at 42°C for 15 minutes, and finally, enzyme inactivation will be performed at 85°C for 5 minutes. Gene expression levels will be determined by the real-time PCR method. The p150 isoform, which is larger in size and has been used in previous studies, will be used. The reaction will be performed in a real-time PCR machine with an initial denaturation step at 95°C for 5 minutes, followed by 40 cycles of 95°C for 5 seconds, 55°C/59°C for 30 seconds (reading).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 50 patients with locally advanced rectal adenocarcinoma scheduled for TNT.: Biopsies will be taken from these 50 patients at the time of diagnosis and after TNT. The relationship between ADAR1 expression levels and TNT response will be investigated.
  Interventions: Genetic: Adenosine deaminase acting on RNA1

INTERVENTIONS:
Genetic: Adenosine deaminase acting on RNA1 — Previous studies have demonstrated that increased ADAR1 expression is associated with poor survival in gastric and metastatic colon cancer. In rectal cancer, however, the relationship between ADAR1 levels and TNT response in locally advanced disease has not been investigated. Another point is that ADAR1 can also be studied using immunohistochemistry; however, its sensitivity and specificity are low, so in our study, RNA will be isolated and analyzed using real-time PCR.

SUMMARY:
Total neoadjuvant therapy (TNT) is currently the standard treatment for locally/locally advanced rectal cancer due to better response and fewer distant metastases. In TNT, sequential chemotherapy (CT) and chemoradiotherapy (CRT) are planned and depending on the treatment response, either surgery is performed or a watch and wait approach is applied. Depending on tumor localization and patient performance status, CT is planned as induction or consolidation. Most of the time, mFOLFOX6 and CAPOX are preferred as CT regimen. In proximal rectal cancer, surgery can be performed without CRT and only after CT. In locally/locally advanced rectal cancer, the aim is to avoid surgery as much as possible or to perform sphincter-sparing surgery if possible. Colonoscopy and pelvic MR at the time of diagnosis are the most important steps in staging, treatment selection and decision making. These two diagnostic methods should be repeated especially for watch and wait decision and for response evaluation after TNT.

ADAR 1 (Adenosine deaminase acting on RNA1) is an RNA editing enzyme that catalyzes the deamination of adenosine to inosine (A-to-I), a dynamic modification that can lead to a diverse transcriptome in a combinatorial manner. A defect in ADAR1-mediated RNA modification results in abnormal regulation of substrates that can affect phenotypic changes in cancer. This phenomenon of over-regulation is seen in many cancers such as colon, liver, lung, breast and esophageal cancers and in many cases promotes tumor progression. In studies, increased ADAR1 expression has been associated with lower survival and worse prognosis, especially in metastatic colon and gastric cancer. ADAR1 is also predicted to increase proliferation through both the AKT pathway and the mTOR pathway and therefore may be targeted in the near future.

ADAR1 expression is monitored by RNA-based real time PCR. In order to demonstrate increased expression, biopsies should be taken from the malignant tissue and the intact tissue of the patient and the biopsy should be stored under -80 C conditions immediately after biopsy to prevent RNA degradation. The tissue will not come into contact with nitrogen or formaldehyde.

In this study, sufficient biopsies from cancerous and intact tissue will be taken from patients with suspected rectal cancer, confirmed by pelvic MRI and consent for participation in the study, and fresh tissue will be stored at -80 C in the genetics laboratory. After the TNT plan is made by the investigators and the treatment is completed, both pelvic MRI and control rectoscopy will be performed for preoperative evaluation. Again, biopsies will be taken from diseased and healthy tissue and ADAR1 expression will be evaluated. The study is planned to include 50 participants and a period of one year is foreseen for tissue procurement/storage.

The investigators' aim in this study will be to determine whether ADAR1 expression level changes after TNT, whether this predicts clinical and pathological response, whether responses change according to the selected CT, whether there is a difference between CT induction-consolidation/RT short or long course, and the relationship between tumor DNA mismatch repair enzyme status and ADAR1 level. The investigators primary endpoint will be the effect of the change in ADAR1 expression level on the response after TNT (ORR). Secondary endpoints will be quality of life, recurrence-free survival (RFS) and overall survival (OS).

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in both sexes, but it ranks second in mortality after lung cancer, with one in ten cancer deaths attributed to colorectal cancer. Total neoadjuvant therapy (TNT) is currently considered the standard of care for the treatment of locally advanced rectal cancer. In this approach, all non-surgical interventions, including multi-agent chemotherapy and concurrent chemoradiotherapy (CRT), are administered prior to surgical resection or the decision to opt for non-operative treatment. Accumulating evidence suggests that TNT improves survival in patients with locally advanced rectal cancer and is expected to reduce distant metastasis through systemic chemotherapy, thereby preventing the onset of micrometastases. TNT has also been associated with improved compliance, reduced toxicity, decreased need for and duration of ileostomy, and improved anal sphincter preservation rates following a watch-and-wait strategy, along with increased complete clinical response. Studies have shown that the rate of pCR in patients receiving TNT therapy is approximately 20-40%. Although numerous randomized controlled trials have evaluated different TNT strategies compared to standard KRT treatment in terms of KRT sequencing, systematic chemotherapy, radiotherapy modality, and TNT intensity, it is known that the TNT approach demonstrates superior survival benefit compared to adjuvant chemotherapy following neoadjuvant KRT. However, TNT theoretically offers several surgical advantages, including an increased likelihood of sphincter-preserving surgery and a reduced need for ileostomy; however, results across studies are inconsistent.

ADAR 1 (Adenosine deaminase acting on RNA1) catalyzes the C6 deamination of adenosine (A) to produce inosine (I) in RNA regions characterized by a double-stranded structure, a process known as adenosine deamination acting on RNA (ATIRE). This process is crucial for altering RNA structures and sequences in both coding and non-coding RNAs, influencing tumor characteristics, tumor stage, drug responses, and patient survival, thereby significantly contributing to cancer progression. The role of ADAR1 in promoting tumorigenesis via the ATIRE pathway is becoming increasingly evident in various cancers, including stomach cancer, esophageal squamous cell carcinoma, breast cancer, hepatocellular carcinoma, and CRC.

ADAR1, ADAR2, and ADAR3 are members of the ADAR family; while ADAR1 and ADAR2 are widely expressed, ADAR3 is primarily expressed in the brain and lacks catalytic activity. ADAR1 contains RNA-binding domains (RBDs) and Zα domains, whereas ADAR2 contains only RBDs. Zα domains enable ADAR1 to bind to newly synthesized RNA and inhibit the activation of pathogenic interferons (IFNs). ADAR1 has two isoforms: an IFN-inducible form (p150) and a constitutively expressed form (p110). It has been found that ADAR1-p110 reduces the chemotactic potential of melanoma cells and promotes immune exclusion . Loss of ADAR1 function results in unregulated RNA accumulation, which can be mistakenly recognized as foreign by RIG-I (Retinoic acid-inducible gene I), thereby triggering its activation and subsequent IFN response. Additionally, DNA released from damaged cells can activate the cGAS (GMP-AMP synthase)-STING (stimulator of interferon genes) pathway, leading to the production of type I IFNs through both pathways. The interaction between ADAR1 and the cGAS-STING and RIG-I pathways highlights a crucial balance in immune regulation. ADAR1's ability to interact with IFNs, regulate IFN production, and its complex roles in cancer therapy, along with its higher expression in MSI-H (microsatellite instability-high) patients, high TMB (tumor mutation burden), PD-1/PDL-1 levels, naive B cells, active memory CD4 T lymphocytes, and M1 macrophage cells, suggests its potential for modulating responses to cancer therapies. A potential mechanism has been proposed whereby increased ADAR1 expression in gastric cancer leads to proliferation and migration of various diseases through the mTOR/p70S6 kinase/S6 ribosomal protein pathway. To investigate the functional relationship between ADAR1 and mTOR signaling, the mTOR kinase inhibitor rapamycin was used to treat gastric cancer cells and observe its effects on ADAR1-overexpressed cell proliferation and migration. The results showed that ADAR1 overexpression significantly promoted cell proliferation and migration as expected, but these effects were significantly attenuated in cells treated with rapamycin. This suggests that rapamycin may block the effects of ADAR1 overexpression on gastric cancer cell growth and migration. These results indicate that the mTOR signaling pathway is important for ADAR1-mediated gastric cancer progression.

Recently, the effect of increased ADAR1 expression on survival in metastatic colon cancer was investigated. Both overall survival (OS) and relapse-free survival (RFS) were found to be significantly reduced in the group with increased ADAR1 expression; however, the study did not include patients with early-stage rectal cancer[20]. For all these reasons, the prognostic value of ADAR1 expression levels and/or changes in locally advanced rectal cancer patients for TNT response will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histological and staging diagnosis of local/locally advanced rectal cancer
* ECOG performance score between 0 and 2
* No contraindications for chemotherapy (CT) and/or radiotherapy (RT)

Exclusion Criteria:

* Those diagnosed with metastatic rectal cancer
* Those suspected of having rectal cancer or patients with a diagnosis of a second primary cancer
* Those who have not signed the informed consent form
* Those with contraindications for chemotherapy (CT) and/or radiation therapy (RT)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced rectal cancer who presented to the medical oncology, radiation oncology, and general surgery clinics of Necmettin Erbakan University Faculty of Medicine Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate according to RECIST 1.1 | From enrollment to the end of treatment at 12 weeks
  Evaluation of target lesions
  Complete Response (CR):
  Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR):
  At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
  Progressive Disease (PD):
  At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD):
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
Recurrence free survival | Disease-free survival is evaluated up to 120 months after the first documented progression or death from any cause (whichever comes first) following surgery or watch and wait decision after TNT.
  Recurrence-free survival refers to the period of time after treatment when a patient remains free of tumor recurrence.
Assessment of Quality of Life | every 3 months for 1 year.
  Quality of life will be assessed using The European Organisation for Research and Treatment of Cancer (EORTC) quality of life (QLQ-C30) questionnaire, which consists of 30 items, every 3 months for 1 year. Higher scores on this quality of life scale are associated with better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Artaç, MD, Study Director — Necmettin Erbakan University Faculty of Medicine, Department of Medical Oncology
Locations (1):
- Necmettin Erbakan University Faculty of Medicine, Departmen of Medical Oncology, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be ready in September 2026 and can be shared within the following year.
Access Criteria: The statistical methods used for objective response rates, survival data, and quality of life outcomes can be reviewed by an independent review.

REFERENCES:
- [Result] Wang Q, Li X, Qi R, Billiar T. RNA Editing, ADAR1, and the Innate Immune Response. Genes (Basel). 2017 Jan 18;8(1):41. doi: 10.3390/genes8010041. PMID 28106799
- [Result] Okugawa Y, Toiyama Y, Shigeyasu K, Yamamoto A, Shigemori T, Yin C, Ichikawa T, Yasuda H, Fujikawa H, Yoshiyama S, Hiro J, Ohi M, Araki T, Kusunoki M, Goel A. Enhanced AZIN1 RNA editing and overexpression of its regulatory enzyme ADAR1 are important prognostic biomarkers in gastric cancer. J Transl Med. 2018 Dec 18;16(1):366. doi: 10.1186/s12967-018-1740-z. PMID 30563560
- [Result] Shigeyasu K, Okugawa Y, Toden S, Miyoshi J, Toiyama Y, Nagasaka T, Takahashi N, Kusunoki M, Takayama T, Yamada Y, Fujiwara T, Chen L, Goel A. AZIN1 RNA editing confers cancer stemness and enhances oncogenic potential in colorectal cancer. JCI Insight. 2018 Jun 21;3(12):e99976. doi: 10.1172/jci.insight.99976. eCollection 2018 Jun 21. PMID 29925690
- [Result] Chan TH, Lin CH, Qi L, Fei J, Li Y, Yong KJ, Liu M, Song Y, Chow RK, Ng VH, Yuan YF, Tenen DG, Guan XY, Chen L. A disrupted RNA editing balance mediated by ADARs (Adenosine DeAminases that act on RNA) in human hepatocellular carcinoma. Gut. 2014 May;63(5):832-43. doi: 10.1136/gutjnl-2012-304037. Epub 2013 Jun 13. PMID 23766440
- [Result] Eisenberg E, Levanon EY. A-to-I RNA editing - immune protector and transcriptome diversifier. Nat Rev Genet. 2018 Aug;19(8):473-490. doi: 10.1038/s41576-018-0006-1. PMID 29692414
- [Result] Chua YJ, Barbachano Y, Cunningham D, Oates JR, Brown G, Wotherspoon A, Tait D, Massey A, Tebbutt NC, Chau I. Neoadjuvant capecitabine and oxaliplatin before chemoradiotherapy and total mesorectal excision in MRI-defined poor-risk rectal cancer: a phase 2 trial. Lancet Oncol. 2010 Mar;11(3):241-8. doi: 10.1016/S1470-2045(09)70381-X. Epub 2010 Jan 25. PMID 20106720
- [Result] Glynne-Jones R, Grainger J, Harrison M, Ostler P, Makris A. Neoadjuvant chemotherapy prior to preoperative chemoradiation or radiation in rectal cancer: should we be more cautious? Br J Cancer. 2006 Feb 13;94(3):363-71. doi: 10.1038/sj.bjc.6602960. PMID 16465172
- [Result] Aref A, Abdalla A. Erratum: Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer: Induction or Consolidation Chemotherapy? J Clin Oncol. 2025 Mar;43(7):898. doi: 10.1200/JCO-25-00095. Epub 2025 Jan 24. No abstract available. PMID 39854654
- See also: ADAR1 in colon cancer — https://pubmed.ncbi.nlm.nih.gov/29925690/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT07108348/Prot_SAP_000.pdf